CLINICAL TRIAL: NCT01951690
Title: Phase II Study of VS-6063, A Focal Adhesion Kinase (FAK) Inhibitor, in Patients With KRAS Mutant Non-Small Cell Lung Cancer
Brief Title: Phase II Study of VS-6063 in Patients With KRAS Mutant Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Verastem, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VS-6063-201
Record Dates: First submitted 2013-09-23; First posted 2013-09-27 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Non Small Cell Lung Cancer; Lung Cancer
Keywords: Focal Adhesion Kinase inhibitor; FAK inhibitor; Cancer Stem Cells; CSC; KRAS mutation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — defactinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VS-6063 (defactinib) (Experimental): Administered orally BID in a 21 day cycle
  Interventions: Drug: defactinib (VS-6063)

INTERVENTIONS:
Drug: defactinib (VS-6063)

SUMMARY:
This is a Phase II, open-label, multicenter, multi cohort, study of VS-6063 (defactinib), a focal adhesion kinase inhibitor, in patients with KRAS mutant non-small cell lung cancer (NSCLC). NSCLC with a KRAS mutation is required for study entry and subjects will be enrolled into 1 of 4 cohorts based on the status of their INK4a/Arf and p53 mutations. The purpose of this study is to demonstrate if VS-6063 (defactinib) improves PFS within each cohort. The safety and tolerability of VS-6063, tumor response rate, progression free survival and overall survival will also be assessed. The pharmacodynamic effects of VS-6063 (defactinib) will be examined in a tumor biopsy and a blood sample.

DETAILED DESCRIPTION:
Eleven subjects will be enrolled into one of four cohorts: Cohort A (KRAS mutation, wild type INK4a/ARF and wildtype p53), Cohort B (KRAS mutation, INK4s/ARF mutation and wild type p53), Cohort C (KRAS mutation, wild type INK4a/ARF and p53 mutation), and Cohort D (KRAS mutation, INK4a/ARF mutation and p53 mutation). If >/= 4 patients demonstrate PFS at 12 weeks in each cohort, an additional 23 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age.
* ECOG (Eastern Cooperative Oncology Group) Performance Score of 0 or 1.
* Histologic or cytologic confirmation of non-small cell lung cancer (NSCLC)
* Molecular characterization of the tumor demonstrating a KRAS mutation by a CLIA-certified assay. Adequate archival tissue, tissue core biopsy specimen, or DNA samples must be available for central testing of INK4a/Arf and p53 if not previously performed by a CLIA certified lab.
* Documented evidence of distant metastasis or locoregional recurrence per required assessments within 28 days prior to starting study therapy.

Note: Histologic confirmation of metastatic disease is not required.

* For patients with brain metastases, the following criteria must be met:

Previously untreated brain metastases that are asymptomatic and not requiring steroids are permitted.

Previously treated brain metastases are permitted if most recent CNS radiographic imaging demonstrates no evidence of CNS disease progression For patients with previously untreated brain metastases, Central Nervous System (CNS) imaging is required at the time of disease imaging throughout treatment.

* At least one measurable disease site per RECIST v1.1.
* Received a minimum of one course of treatment that included at least one platinum-based chemotherapy doublet for metastatic or locally recurrent disease.
* Adequate hematologic function including ANC ≥ 1200/mm3, Hemoglobin ≥ 9 g/dL (transfusion is permitted), and platelets ≥ 100,000/mm3.
* Adequate hepatic function including ALT ≤ 2.5 x upper limit of normal (ULN) if liver metastasis is NOT present or ≤ 5 x ULN if liver metastasis is present, and total bilirubin ≤ 1.5 x ULN.
* QTc (corrected QT) interval < 480 msec.

Exclusion Criteria:

* Presence of an activating EGFR (epidermal growth factor receptor) mutation or ALK (anaplastic lymphoma kinase) translocation in the tumor.
* Radiotherapy (RT) completed within 14 days prior to the first dose of study therapy.
* Known impairment of gastrointestinal function that would alter drug absorption.
* Leptomeningeal metastasis.
* Symptomatic or untreated brain metastases or spinal cord compression or any of these conditions requiring chronic steroids to control symptoms.
* History or evidence of cardiac risk
* Known history of malignant hypertension (severe hypertension >180/120 mmHg with end organ involvement.
* Another active concurrent malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Demonstrate that VS-6063 (defactinib), will improve PFS at 12 weeks (PFS12) within each cohort. | From baseline through 12 weeks of treatment

SECONDARY OUTCOMES:
Evaluate the response rate (RR) | Every 6 weeks from baseline through the end of treatment, an expected average of 4 months
  RR is measured as the best overall response using Response Evaluation Criteria In Solid Tumors (RECIST), version 1.1.
Evaluate progression free survival | From the date of first treatment to the date of progression including death from any cause, expected average at least 4 months
  PFS will be estimated in each cohort using Kaplan-Meier product limit estimates.
Evaluate Overall Survival (OS) | OS will be calculated from the date of first treatment to the date of death from any cause, expected average of at least 12 months. Patients who did not experience death will be censored at the last follow-up time.
  OS in each cohort will be estimated using Kaplan-Meier product limit estimates.

OTHER OUTCOMES:
Evaluation of the association between pharmacodynamic (PD) biomarkers and clinical outcomes (response rate, progression-free survival and overall survival) | Baseline PD biomarkers will be associated with the RR (collected every 6 weeks) and PFS, both with expected average of 4 months from first treatment to progression, and OS (expected average of 12 months from first treatment to date of death)
Evaluate the safety and tolerability of VS-6063 (defactinib) | From start of treatment to end of treatment, an expected average of 4 months
  Adverse events (AEs) include the incidences of all treatment-emergent AEs (TEAEs) and all Serious Adverse Events (SAEs); by severity, relationship to study drug, and discontinuation of patients from study therapy due to AEs and due to deaths. Safety endpoints for AEs, clinical laboratory tests, vital signs, ECGs and physical examinations will be summarized using descriptive statistics as determined based on CTCAE (Common Toxicity Criteria for Adverse Effects) 4.03

CONTACTS AND LOCATIONS:
Overall Officials: David E Gerber, M.D., Principal Investigator — University of Texas Southwestern Medical Center
Locations (9):
- United States (9):
  - University of Colorado Cancer Center, Anschutz Medical Campus, Denver, Colorado
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Johns Hopkins Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Knight Cancer Institute, Oregon Health and Science University, Portland, Oregon
  - University of Pittsburgh Medical Center Cancer Center, Pittsburgh, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas

REFERENCES:
- [Derived] Shimizu T, Fukuoka K, Takeda M, Iwasa T, Yoshida T, Horobin J, Keegan M, Vaickus L, Chavan A, Padval M, Nakagawa K. A first-in-Asian phase 1 study to evaluate safety, pharmacokinetics and clinical activity of VS-6063, a focal adhesion kinase (FAK) inhibitor in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2016 May;77(5):997-1003. doi: 10.1007/s00280-016-3010-1. Epub 2016 Mar 30. PMID 27025608